CLINICAL TRIAL: NCT01331811
Title: Improving Diagnosis of Tuberculosis in HIV Infected Children in Asia (Cambodia, Vietnam) and Africa (Burkina Faso, Cameroon) ANRS 12229 PAANTHER 01 (Pediatric Asian African Network for Tuberculosis and HIV Research)
Brief Title: Improving Diagnosis of Tuberculosis in HIV Infected Children in Asia (Cambodia, Vietnam)and Africa (Burkina Faso, Cameroon)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut Pasteur, Cambodia (Other); National Pediatric Hospital, Cambodia (Unknown); Angkor Hospital for Children (Other); Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam (Other); Pediatric Hospital Nhi Dong 1, Ho Chi Minh City, Vietnam (Unknown); Number 2 Children's Hospital, Ho Chi Minh City (Other); Hôpital Necker-Enfants Malades, Paris, France (Unknown); Groupe Hospitalier Pitie-Salpetriere (Other); CHRU Arnaud de Villeveuve, Montpellier, France (Unknown); IRD, Yaounde, Cameroon (Unknown); Fondation Chantal Biya,Yaounde, Cameroon (Unknown); CHU Sourô Sanou, Bobo Dioulasso, Burkina Faso (Unknown); Centre Muraz (Other); Centre Pasteur du Cameroun (Other); Centre Hospitalier D'essos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANRS12229 PAANTHER 01
Record Dates: First submitted 2011-04-04; First posted 2011-04-08 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: HIV; Tuberculosis; Pediatrics
Keywords: HIV; Tuberculosis; Diagnosis; Pediatrics; Asia; Africa
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Development of a diagnosis algorithm — At entry in the study, HIV infected children with suspected tuberculosis will undergo a complete evaluation including:
  * interview on anamnesis
  * clinical examination
  * evaluation of HIV infection stage
  * hematology and biochemistry tests
  * CD4 count
  * HIV viral load
  * IGRA
  * chest radiograph
  * Abdominal ultrasonograph to detect abdominal lymphadenopathy
  * Tuberculin skin test
  * gastric aspirates, sputum and string tests according to the age of children
  * nasopharyngeal aspirate
  * stool sample
  * lymph node fine needle aspirate or other specimen collection if applicable
  Diagnosis and treatment of all participating children will be done according to national guidelines. The children will be followed-up for 6 months until the end of their anti-TB treatment. For the analysis of data and the validation of the algorithm, children will be randomized into 2 groups. Data from Group I will be used to develop the algorithm; data from Group II will be used to validate it.

SUMMARY:
Childhood tuberculosis (TB) accounts for 11% of the total 9 million annual TB cases and the difficulty of its diagnosis is increased in case of HIV infection in children.

The aim of this study is to improve TB diagnosis in HIV-infected children by developing a new diagnostic algorithm incorporating new tools available such as:

* interferon gamma release assays (IGRAs), as alternative to the tuberculin skin test
* alternative specimen collection methods such as string test (or Enterotest (R)), nasopharyngeal aspirates and stools samples, as alternatives to gastric aspirate
* the Xpert MTB/RIF assay

ELIGIBILITY:
Inclusion Criteria:

* children aged from 0 to 13 years
* confirmed HIV infection
* suspicion of tuberculosis
* informed consent signed by at least one parent or guardian
* on ARVs or not

Exclusion Criteria:

* history of anti TB treatment started in the past 2 years
* on going tuberculosis treatment
* Suspicion of exclusive extra-thoracic tuberculosis

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 441 (Actual)
Dates: Start 2011-04; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Tuberculosis diagnostic algorithm | 3 years
  Development of an effective diagnostic algorithm for pediatric tuberculosis after evaluating the following diagnostic tests and sampling methods:
  * Clinical examination
  * Chest X-rays
  * Abdominal ultrasound
  * IGRAs
  * Xpert MTB/RIF
  * Gastric aspirate
  * String test
  * Nasopharyngeal aspirate
  * Stools sample
  * Sputum samples

SECONDARY OUTCOMES:
Evaluation of the QuantiFERON(R)-TB Gold In-Tube | 6 months
  Evaluation of the sensitivity, specificity, positive and negative predictive values of an in-vitro Interferon Gamma Release (IGRAs) : the QuantiFERON(R)-TB Gold iIn-Tube, for the diagnosis of TB in HIV infected children
Comparison of two in-vitro IGRAs | 6 months
  Comparison of the performances of two in-vitro IGRAs: the QauntiFERON(R)-TB Gold In-Tube and the T.SPOT-TB(R), for the diagnosis of tuberculosis in a sub-group of HIV infected children.
Percentage of TB diagnosis sampling procedures actually performed | 6 months
  To assess the feasibility of the following TB sampling procedures:
  * the string test
  * the nasopharyngeal aspirate
  * stool sample
Evaluation of the morbidity (IRIS, drug toxicity and other opportunistic infections) and mortality in TB-HIV co-infected children | at 6 month of TB treatment
Specificity and sensibility of TB diagnosis sampling procedures compared to TB diagnosis gold standard (sputum or gastric aspirate culture) | 6 months
  To assess the performance of the following TB sampling procedures:
  * the string test
  * the nasopharyngeal aspirate
  * stools sample
Evaluation of the Xpert MTB/RIF assay | 6 months
  Evaluate the sensitivity, specificity, positive and negative predictive values of the Xpert MTB/RIF assay
Comparison of the Xpert MTB/RIF test to the gold standard (culture of gastric aspirates or sputum) | 6 months
Comparison of the performance Xpert MTB/RIF assay on sampling methods other than the reference method (gastric aspirate and sputum) | 6 months
  Evaluation of the Xpert MTB/RIF assay on the following sampling methods:
  * String test
  * Nasopharyngeal aspirates
  * Stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Marcy, MD, Study Chair — Institut Pasteur in Cambodia, Phnom Penh, Cambodia; Vibol Ung, MD, Study Chair — National Pediatric Hospital, Phnom Penh, Cambodia
Locations (8):
- CHU Sourô Sanou, Bobo-Dioulasso, Burkina Faso
- Cambodia (2):
  - National Pediatric Hospital, Phnom Penh
  - Angkor Hospital for Children, Siem Reap
- Cameroon (2):
  - Centre Hospitalier d'Essos, Yaoundé
  - Centre Mère Enfant Chantal Biya, Yaoundé
- Vietnam (3):
  - Pediatric Hospital Nhi Dong 1, Ho Chi Minh City
  - Pediatric Hospital Nhi Dong 2, Ho Chi Minh City
  - Pham Ngoc Thach Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Marcy O, Borand L, Ung V, Msellati P, Tejiokem M, Huu KT, Do Chau V, Ngoc Tran D, Ateba-Ndongo F, Tetang-Ndiang S, Nacro B, Sanogo B, Neou L, Goyet S, Dim B, Pean P, Quillet C, Fournier I, Berteloot L, Carcelain G, Godreuil S, Blanche S, Delacourt C; ANRS 12229 PAANTHER 01 STUDY GROUP. A Treatment-Decision Score for HIV-Infected Children With Suspected Tuberculosis. Pediatrics. 2019 Sep;144(3):e20182065. doi: 10.1542/peds.2018-2065. PMID 31455612
- [Derived] Borand L, de Lauzanne A, Nguyen NL, Cheng S, Pham TH, Eyangoh S, Ouedraogo AS, Ung V, Msellati P, Tejiokem M, Nacro B, Inghammar M, Dim B, Delacourt C, Godreuil S, Blanche S, Marcy O; Pediatric Asian African Network for Tuberculosis and HIV Research (PAANTHER) Study Group. Isolation of Nontuberculous Mycobacteria in Southeast Asian and African Human Immunodeficiency Virus-infected Children With Suspected Tuberculosis. Clin Infect Dis. 2019 May 2;68(10):1750-1753. doi: 10.1093/cid/ciy897. PMID 30689814
- [Derived] Marcy O, Tejiokem M, Msellati P, Truong Huu K, Do Chau V, Tran Ngoc D, Nacro B, Ateba-Ndongo F, Tetang-Ndiang S, Ung V, Dim B, Neou L, Berteloot L, Borand L, Delacourt C, Blanche S; ANRS 12229 PAANTHER 01 Study Group. Mortality and its determinants in antiretroviral treatment-naive HIV-infected children with suspected tuberculosis: an observational cohort study. Lancet HIV. 2018 Feb;5(2):e87-e95. doi: 10.1016/S2352-3018(17)30206-0. Epub 2017 Nov 23. PMID 29174612
- [Derived] Marcy O, Ung V, Goyet S, Borand L, Msellati P, Tejiokem M, Nguyen Thi NL, Nacro B, Cheng S, Eyangoh S, Pham TH, Ouedraogo AS, Tarantola A, Godreuil S, Blanche S, Delacourt C. Performance of Xpert MTB/RIF and Alternative Specimen Collection Methods for the Diagnosis of Tuberculosis in HIV-Infected Children. Clin Infect Dis. 2016 May 1;62(9):1161-1168. doi: 10.1093/cid/ciw036. Epub 2016 Feb 7. PMID 26908804